CLINICAL TRIAL: NCT03687125
Title: Phase 1/2 Open-label Trial of Tinostamustine Conditioning and Autologous Stem Cell Transplantation for Salvage Treatment in Relapsed / Refractory Multiple Myeloma (TITANIUM 1)
Brief Title: Tinostamustine Conditioning and Autologous Stem Cell
Acronym: TITANIUM1
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision based on adverse events limiting administration of higher doses required to achieve myeoblative conditioning necessary in this population
Sponsor: Mundipharma-EDO GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EDO-S101-1004; 2018-001907-35 (EudraCT Number)
Record Dates: First submitted 2018-08-29; First posted 2018-09-27 (Actual); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-05

CONDITIONS: Multiple Myeloma in Relapse; Multiple Myeloma Progression; Multiple Myeloma With Failed Remission
MeSH Terms: interventions — tinostamustine

STUDY DESIGN:
Intervention Model Description: Phase 1 Does escalation followed by Phase 2 Expansion at MTD
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tinostamustine 180 mg/m^2 (Experimental): Participants received single dose of tinostamustine 180 milligrams per meter square (mg/m^2) intravenous (IV) injection on Day -1 followed by autologous stem cell transplantation (ASCT) on Day 1.
  Interventions: Drug: Tinostamustine; Procedure: Autologous Stem Cell Transplant (ASCT)
- Tinostamustine 220 mg/m^2 (Experimental): Participants received single dose of tinostamustine 220 mg/m^2 IV injection on Day -1 followed by ASCT on Day 1.
  Interventions: Drug: Tinostamustine; Procedure: Autologous Stem Cell Transplant (ASCT)

INTERVENTIONS:
Drug: Tinostamustine — Participants received tinostamustine IV injection.
Procedure: Autologous Stem Cell Transplant (ASCT) — Undergo autologous stem cell transplant

SUMMARY:
Phase 1

The primary objectives of Phase 1 of this study are to:

* Establish the safety, toxicity, and maximum tolerated dose (MTD) of the tinostamustine conditioning regimen.
* Identify the recommended Phase 2 dose (RP2D) of tinostamustine for use in the Phase 2 portion of the study.

The secondary objective of Phase 1 of this study is to:

- Investigate the pharmacokinetics (PK) of tinostamustine.

DETAILED DESCRIPTION:
Study Design (Methodology):

This is a 2-part, international, multi-center, open-label study of salvage treatment with tinostamustine conditioning followed by ASCT in participants with relapsed/ refractory multiple myeloma (MM). (ASCT is defined as salvage if the participant had already received a prior ASCT and undergoes a second ASCT after evidence of progressive disease [PD].) Phase 1 of the study employs a standard 3+3 dose escalation design with the objective of defining the dose limiting toxicities (DLTs) of the tinostamustine conditioning regimen and defining the MTD and RP2D for use in the Phase 2 portion of the study.

The Safety Review Committee can make a decision to stop dose escalation or explore intermediary doses at any time. The total dose of tinostamustine will be administered on Day -1. Phase 2 of the study employs a 2-step sequential design (Simon, 1989). In Stage 1 of Phase 2, up to 31 participants initially will be enrolled. If lesser than or equal to (<=) 25 participants of these initial 31 participants experience a response, then no additional participants will be enrolled. However, if greater than (>) 25 participants in Stage 1 of Phase 2 experience a response, then enrollment in this cohort will continue, with up to 71 participants enrolled. In Phase 2 of the study, all participants will receive tinostamustine at the RP2D administered in Phase 1 according to the same schedule. After provision of written informed consent, participants will be screened for study eligibility within 28 days before Day 1 (the day of ASCT). Participants who have a minimum of 2×106 CD34+ cells/kg cryopreserved and are otherwise determined to be eligible, based on screening assessments, will be enrolled and receive the tinostamustine conditioning regimen. The tinostamustine dose will be administered 24 hours pre-ASCT (i.e., Day -1). On Day 1, ASCs will be administered intravenously (IV) according to standard institutional practice. Participants will receive supportive measures (including growth factor support post-ASCT, antimicrobial prophylaxis, red blood cell and platelet transfusion, and treatment for neutropenic fever) according to standard institutional practice.

ELIGIBILITY:
Inclusion Criteria:

1. Participants has Multiple Myeloma (MM) and:

   a. Has received prior ASCT after standard first-line induction treatment. b. Has evidence of progressive disease (PD), with progression-free interval greater than or equal to (>=) 6 months in Phase 1 >= 18 months in Phase 2.
   * Progression Free Interval is defined as the time from date of ASCT to PD. c. Received treatment with lesser than or equal to (<=) 3 prior lines of therapy.
   * A line of therapy is defined as 1 or more cycles of a planned treatment program. When participants have undergone sequential phases of treatment without intervening progression, such as induction, collection of peripheral blood stem cells (PBSCs), transplantation and consolidation/maintenance, this is considered to be 1 line of treatment. A new line of therapy is initiated as a result of PD or relapse.
2. Complete response (CR), very good partial response (VGPR), partial response (PR), or minimal response (MR) to salvage chemotherapy, as determined by the International Myeloma Working Group (IMWG) criteria.
3. Is, in the Investigator's opinion, a candidate for consolidation therapy with tinostamustine followed by ASCT. (Note that participants planned to receive tandem ASCT are not eligible for the Phase 1 portion of the study.)
4. Has available autologous peripheral blood stem cell (PBSC) product with CD34 cell dose >= 2×106 cells/kg. The product could be from a collection prior to first ASCT or later second collection. (Note that, although not required, in Phase 1, the Investigator should consider enrolling participant with a large number of available PBSCs to permit subsequent ASCT, as participants in Stage 1 may received a dose lower than that determined to be effective.)
5. Age 18-75 years.
6. Eastern Cooperative Oncology Group (ECOG) performance status score lesser than (<) 3 at Screening.
7. Creatinine clearance >= 40 milliliter per minute (mL/min), as determined by a local laboratory using the Cockcroft-Gault equation within 28 days before ASCT.
8. Left ventricular ejection fraction (LVEF) >= 40 percent (%) within 28 days before ASCT.
9. Adequate pulmonary function, defined as forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), and carbon monoxide diffusing capacity (DLCO) greater than (>) 50% predicted within 28 days before ASCT.
10. Adequate liver function, as defined by an alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <= 2.5 × the upper limit of normal (ULN) and bilirubin <= 1.5 × ULN within 28 days before ASCT.
11. Potassium within the local laboratory's normal range. (Potassium supplementation is permissible.)

Exclusion Criteria:

Participants meeting any of the following criteria are not eligible for study entry:

1. History of central nervous system (CNS) disease involvement.
2. Primary or secondary plasma cell leukemia at any time point prior to transplant.
3. Myocardial infarction (MI) or stroke within 6 months before Screening.
4. Uncontrolled acute infection.
5. Hematopoietic cell transplantation-comorbidity index (HCT-CI) > 6 points.
6. Concurrent malignant disease with the exception of treated basalioma/spinalioma of the skin or early-stage cervix carcinoma, or early-stage prostate cancer. Previous treatment for other malignancies (not listed above) must have been terminated at least 24 months before registration and no evidence of active disease shall be documented since then.
7. Major coagulopathy or bleeding disorder.
8. Other serious medical condition that could potentially interfere with the completion of treatment according to this protocol or that would impair tolerance to therapy or prolong hematological recovery.
9. Lack of cooperation to allow study treatment as outlined in this protocol.
10. Pregnancy or lactating female participants.
11. The use of any anti-cancer investigational agents within 21 days prior to the expected start of trial treatment and interval of 14 days to last administration of salvage treatment.
12. Receiving treatment with drugs known to prolong the QT/QTc interval.
13. QTc interval (Fridericia's formula) > 450 millisecond (msec), based on the mean of triplicate Screening 12-lead electrocardiograms (ECGs).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parameswaran Hari, MD, Study Chair — Study Chair; Dagmar Hess, Study Chair — 2nd Study Chair
Locations (12):
- United States (7):
  - University of Alabama, Birmingham, Alabama
  - University of Kansas Medical Center Kansas City, Kansas City, Kansas
  - Memorial Sloan Kettering Cancer Centre, New York, New York
  - Carolinas Healthcare System, Charlotte, North Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Froedtert & Medical College of Wisconsin, Cancer Center - Froedtert Hospital, Milwaukee, Wisconsin
- Oslo Myeloma Center, Oslo University Hospital, Oslo, Norway
- Switzerland (4):
  - Universitatsspital Basel, Basel
  - Universitatsspital Bern, Bern
  - Department of Clinical Research Oncology/Hematology, Kantonsspital St. Gallen, Sankt Gallen
  - University Hospital Zurich, Zurich

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 3 centers in the United States between 15 October 2018 and 17 April 2019.
Pre-assignment Details: A total of 6 participants were enrolled and received study drug in Phase 1. Study was early terminated during Phase 1 due to sponsor decision on 17 April 2019 (adverse events limited administration of higher doses required to achieve myeoblative conditioning necessary in this population). Hence, no participants were enrolled in Phase 2 and efficacy analysis were not performed in the both Phase 1 and 2.
Period: Overall Study
Arm/Group | Tinostamustine 180 mg/m^2 | Tinostamustine 220 mg/m^2
Started | 3 | 3
Completed | 0 | 2
Not Completed | 3 | 1
Not completed — Progressive Disease | 2 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received tinostamustine.
Groups:
- Tinostamustine 180 mg/m^2: Participants received single dose of tinostamustine 180 mg/m^2 IV injection followed by autologous stem cell transplantation (ASCT) on Day 1.
- Tinostamustine 220 mg/m^2: Participants received single dose of tinostamustine 220 mg/m^2 IV injection followed by ASCT on Day 1.
- Total: Total of all reporting groups
Arm/Group | Tinostamustine 180 mg/m^2 | Tinostamustine 220 mg/m^2 | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.3 (7.37) | 61.3 (11.02) | 62.3 (8.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White/Caucasian | 2 | 1 | 3
  Race: Black | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Phase 2: Objective Response Rate (ORR) Based on International Myeloma Working Group (IMWG) Response Criteria
Description: ORR was defined as the participants with a complete response (CR) or very good partial response (VGPR) or partial response (PR) as determined by IMWG Response Criteria. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (target/non target) must have reduction in short axis to less than (<) 10 mm; PR was defined as at least 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum longest diameter; VGPR was defined as a >90% reduction in serum IgM levels from baseline.
Time Frame: at Day 100 post-autologous stem cell transplant (ASCT)
Population: The study was early terminated on 17 April 2019, due to safety signals during Phase 1, participants were not enrolled in Phase 2. Hence, no efficacy analysis were analyzed or collected in this study.
Groups:
- Tinostamustine 180 mg/m^2: Participants received single dose of tinostamustine 180 mg/m^2 IV injection on Day -1 followed by ASCT on Day 1.
Arm/Group | Tinostamustine 180 mg/m^2 | Tinostamustine 220 mg/m^2
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Phase 1: Number of Participants With Dose Limiting Toxicities (DLT)
Description: DLT was defined as at least possibly related to tinostamustine based on common terminology criteria for adverse events 4.03 (CTCAE 4.03): (1) delayed engraftment (greater than [>] 30 days after ASCT) where subject has not met criteria for both neutrophil (first of 3 consecutive days with ANC > 0.5×10^9/liter [L]) and platelet (plt) engraftment (first of 3 consecutive days of plt count > 20×10^9/L without plt transfusion in prior 7 days) (2) QTcF > 500 millisecond (msec) or > 60 msec increase from baseline with duration of > 30 minutes or greater than or equal to (>=) Grade 3 QTcF interval prolongation with ventricular arrhythmia (3) Grade 4 non-hematologic toxicity (4) Grade 3 non-hematologic toxicity related to treatment, except: nausea, emesis, diarrhea, fatigue, dehydration, glucose intolerance, skin rash with treatment, fever (> 40C for >= 24 hours), infection, dyspnea, hypoxia, pneumonitis, pain, dysphagia, oral mucositis, anorexia, flu-like or engraftment syndrome, weight.
Time Frame: Phase 1: From Day -1 up to 30 Days post-ASCT
Population: Safety population included all participants who received tinostamustine. The study was early terminated on 17 April 2019, due to safety signals during Phase 1, participants were not enrolled in Phase 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Tinostamustine 180 mg/m^2 | Tinostamustine 220 mg/m^2
Number analyzed (Participants) | 3 | 3
Participants | 0 | 0

3. Secondary Outcome: Phase 1 and 2: Objective Response Rate (ORR) for Participants Treated at the Recommended Phase 2 Dose (RP2D)
Description: ORR for participants who achieved CR, minimal residual disease negativity (MRD-N), was determined by next generation flow cytometry according to the IMWG Criteria.
Time Frame: at Day 100 post ASCT
Population: as for outcome 1
Arm/Group | Tinostamustine 180 mg/m^2 | Tinostamustine 220 mg/m^2
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Phase 1 and 2: Number of Participants With Neutrophil and Platelet Engraftment Failure
Description: Neutrophil engraftment was defined as the first of 3 consecutive days with absolute neutrophil count (ANC) >0.5 × 10 ^9/L. Platelet engraftment was defined as the first of 3 consecutive days of platelet count >20 × 10 ^9/L without platelet transfusion in the prior 7 days. Number of participants with neutrophil and platelet engraftment failure was reported.
Time Frame: up to 6 months
Population: The study was early terminated on 17 April 2019, due to safety signals during Phase 1. Hence, data for this outcome measure was not collected as planned, analyzed and reported at specific time point.
Arm/Group | Tinostamustine 180 mg/m^2 | Tinostamustine 220 mg/m^2
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Phase 1 and 2: Duration of Cytopenia
Description: Duration of cytopenia i.e ANC <= 0.5×10^9/L, and platelet count <= 20×10^9/L.
Time Frame: Up to 6 months
Population: as for outcome 4
Arm/Group | Tinostamustine 180 mg/m^2 | Tinostamustine 220 mg/m^2
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Phase 1 and 2: Number of Participants With Treatment Related Mortality (TRM)
Description: Number of participants with treatment related mortality was reported.
Time Frame: Up to 6 months
Population: as for outcome 4
Arm/Group | Tinostamustine 180 mg/m^2 | Tinostamustine 220 mg/m^2
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Phase 1 and 2: Number of Participants With Transplant-related Non-hematologic Grade 3 Toxicity
Description: Transplant-related non-hematologic grade 3 toxicity was defined by CTCAE 4.03 stratified by hematopoietic cell transplantation comorbidity index (HCT-CI). HCT-CI is a validated comorbidity index that comprises 17 different categories of organ dysfunction. Positive findings are summated into a total score. The HCT-CI provides information with regard to the overall as well as non-relapse mortality risk a patient is likely to experience after stem cell transplantation (SCT).
Time Frame: Up to 6 months
Population: as for outcome 4
Arm/Group | Tinostamustine 180 mg/m^2 | Tinostamustine 220 mg/m^2
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Phase 1 and 2: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. Serious adverse event (SAE) was defined as AE resulting in any of the following outcomes deemed significant for any other reason: death, was life-threatening (participant was at immediate risk of death from event as it occurred), requires in-patient hospitalization (formal admission to a hospital for medical reasons) or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect. TEAE was defined as an adverse event that started on or after the first dose of tinostamustine through Day 107, or after the end of the study if thought to be related to study drug.
Time Frame: From first dose of tinostamustine up to end of study (up to 6 months)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tinostamustine 180 mg/m^2 | Tinostamustine 220 mg/m^2
Number analyzed (Participants) | 3 | 3
Participants
  Participants with TEAEs | 3 | 3
  Participants with TESAEs | 1 | 2

9. Secondary Outcome: Phase 1 and 2: Change From Baseline in Hematology Parameters
Description: Hematology parameters assessment included white blood cell (WBC) count and differential (lymphocytes, monocytes, basophils, eosinophils, neutrophils), red blood cell (RBC) count, hematocrit, hemoglobin, and platelet count. Change From baseline in hematology parameters at Day 30 were reported.
Time Frame: Baseline (Day -1), Day 30
Population: as for outcome 4
Arm/Group | Tinostamustine 180 mg/m^2 | Tinostamustine 220 mg/m^2
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Phase 1 and 2: Change From Baseline in Clinical Serum Chemistry Tests: Electrolytes
Description: Clinical serum chemistry tests included electrolytes i.e. bicarbonate, calcium, magnesium, chloride, glucose, phosphate, potassium, and sodium. Change from baseline in clinical serum chemistry tests i.e. electrolytes at Day 100 were reported.
Time Frame: Baseline (Day -1), Day 100
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Tinostamustine 180 mg/m^2 | Tinostamustine 220 mg/m^2
Number analyzed (Participants) | 3 | 3
millimoles per liter (mmol/L)
  Bicarbonate: Change at Day 100 | -0.3 (1.53) | -0.7 (1.15)
  Calcium: Change at Day 100 | 0.0667 (0.12332) | 0.1167 (0.07638)
  Chloride: Change at Day 100 | -2.3 (4.04) | -0.3 (1.53)
  Glucose: Change at Day 100 | -3.3121 (4.01991) | -0.7771 (2.69209)
  Magnesium: Change at Day 100 | -0.0274 (0.09501) | -0.0274 (0.04750)
  Phosphate: Change at Day 100 | -0.0969 (0.26439) | -0.2046 (0.29308)
  Potassium: Change at Day 100 | 0.20 (0.265) | 0.10 (0.361)
  Sodium: Change at Day 100 | -2.0 (3.61) | -1.3 (1.15)

11. Secondary Outcome: Phase 1 and 2: Change From Baseline in Clinical Serum Chemistry Tests: Liver Function Parameters
Description: Clinical serum chemistry tests included liver function parameters i.e. Alanine aminotransferase (ALT), Alkaline phosphatase (ALP), Aspartate aminotransferase, (AST) and Lactate dehydrogenase. Change from baseline in clinical serum chemistry tests i.e. liver function parameters at Day 100 were reported.
Time Frame: Baseline (Day -1), Day 100
Population: Safety population included all participants who received tinostamustine. The study was early terminated on 17 April 2019, due to safety signals during Phase 1, participants were not enrolled in Phase 2. Here, number analyzed refers to the number of participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Tinostamustine 180 mg/m^2 | Tinostamustine 220 mg/m^2
Number analyzed (Participants) | 3 | 3
units per liter (U/L)
  ALT: Change at Day 100 | 4.0 (1.73) | 0.3 (3.06)
  ALP: Change at Day 100 | 10.7 (6.81) | 14.7 (5.13)
  AST: Change at Day 100 | 3.0 (1.00) | 2.0 (4.36)
  Lactate dehydrogenase: Change at Day 100: number analyzed (Participants) | 2 | 2
  Lactate dehydrogenase: Change at Day 100 | -21.0 (11.31) | 4.0 (2.83)

12. Secondary Outcome: Phase 1 and 2: Change From Baseline in Clinical Serum Chemistry Tests: Renal Function Parameters
Description: Clinical serum chemistry tests included renal function parameters i.e. creatinine and bilirubin. Change from baseline in clinical serum chemistry tests i.e. renal function parameters at Day 100 were reported.
Time Frame: Baseline (Day -1), Day 100
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Tinostamustine 180 mg/m^2 | Tinostamustine 220 mg/m^2
Number analyzed (Participants) | 3 | 3
millimoles per liter (mmol/L)
  Creatinine: Change at Day 100 | 14.1440 (18.71075) | 25.6360 (8.43282)
  Bilirubin: Change at Day 100 | -1.710 (3.4200) | -3.420 (6.1655)
  Direct Bilirubin: Change at Day 100: number analyzed (Participants) | 2 | 1
  Direct Bilirubin: Change at Day 100 | 0.855 (1.2092) | -3.420 (NA) — NA indicates that standard deviation was not estimated for single participant.
  Indirect Bilirubin: Change at Day 100: number analyzed (Participants) | 2 | 1
  Indirect Bilirubin: Change at Day 100 | 0.855 (1.2092) | -6.840 (NA) — NA indicates that standard deviation was not estimated for single participant.

13. Secondary Outcome: Phase 1 and 2: Change From Baseline in Clinical Serum Chemistry Tests: Total Protein
Description: Clinical serum chemistry tests included total protein. Change from baseline in clinical serum chemistry tests i.e. total protein at Day 100 were reported.
Time Frame: Baseline (Day -1), Day 100
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | Tinostamustine 180 mg/m^2 | Tinostamustine 220 mg/m^2
Number analyzed (Participants) | 3 | 3
gram per liter (g/L) | 13.67 (11.372) | 30.13 (32.309)

14. Secondary Outcome: Phase 1 and 2: Time to Reach Maximum Plasma Concentration (Tmax) of Tinostamustine and Its Metabolites
Description: Tmax was defined as time to reach maximum plasma concentration. Tinostamustine (EDO-S101) and its metabolites included M2-EDO-S101 and M8-EDO-S101.
Time Frame: Pre-infusion, 0.50, 0.75, 1, 3, 6, 24, 48 hours post-infusion
Population: Pharmacokinetic (PK) population included all participants in the safety population with at least one quantifiable pre-dose and one quantifiable post-dose PK plasma concentration. The study was early terminated on 17 April 2019, due to safety signals during Phase 1, participants were not enrolled in Phase 2.
Measure: Median (Full Range); unit: hours
Arm/Group | Tinostamustine 180 mg/m^2 | Tinostamustine 220 mg/m^2
Number analyzed (Participants) | 3 | 3
hours
  EDO-S101 | 0.75 [0.50 to 0.75] | 0.75 [0.50 to 0.75]
  M2-EDO-S101 | 1.00 [1.00 to 1.00] | 1.00 [0.75 to 3.00]
  M8-EDO-S101 | 0.75 [0.50 to 0.75] | 1.00 [0.50 to 1.00]

15. Secondary Outcome: Phase 1 and 2: Maximum Observed Plasma Concentration (Cmax) of Tinostamustine and Its Metabolites
Description: Cmax was defined as maximum observed plasma concentration. Tinostamustine (EDO-S101) and its metabolites included M2-EDO-S101 and M8-EDO-S101.
Time Frame: Pre-infusion, 0.50, 0.75, 1, 3, 6, 24, 48 hours post-infusion
Population: PK population included all participants in the safety population with at least one quantifiable pre-dose and one quantifiable post-dose PK plasma concentration. The study was early terminated on 17 April 2019, due to safety signals during Phase 1, participants were not enrolled in Phase 2.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Tinostamustine 180 mg/m^2 | Tinostamustine 220 mg/m^2
Number analyzed (Participants) | 3 | 3
nanogram per milliliter (ng/mL)
  EDO-S101 | 2270 (910) | 3070 (1320)
  M2-EDO-S101 | 2.85 (1.45) | 2.23 (0.633)
  M8-EDO-S101 | 52.4 (4.58) | 60.4 (11.5)

16. Secondary Outcome: Phase 1 and 2: Area Under the Concentration-time Curve From Time Zero to the Last Measurable Concentration (AUC0-t) of Tinostamustine and Its Metabolites
Description: AUC0-t was defined as area under the concentration-time curve from time zero to the last measurable concentration. Tinostamustine (EDO-S101) and its metabolites included M2-EDO-S101 and M8-EDO-S101.
Time Frame: Pre-infusion, 0.50, 0.75, 1, 3, 6, 24, 48 hours post-infusion
Population: PK population included all participants in the safety population with at least one quantifiable pre-dose and one quantifiable post-dose PK plasma concentration. The study was early terminated on 17 April 2019, due to safety signals during Phase 1, participants were not enrolled in Phase 2. Here, number analyzed refers to the number of participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Tinostamustine 180 mg/m^2 | Tinostamustine 220 mg/m^2
Number analyzed (Participants) | 3 | 3
hour*nanogram per milliliter (h*ng/mL)
  EDO-S101 | 2858.44 (1475.82) | 4922.66 (2056.86)
  M2-EDO-S101: number analyzed (Participants) | 2 | 3
  M2-EDO-S101 | NA (NA) — Mean and Standard Deviation (SD) was not calculated as data were available for only two participants. | 6.65 (3.75)
  M8-EDO-S101 | 60.42 (20.36) | 100.75 (20.01)

17. Secondary Outcome: Phase 1 and 2: Area Under the Concentration-time Curve From Time Zero to 12 Hours (AUC0-12h) of Tinostamustine and Its Metabolites
Description: AUC0-12h was defined as area under the concentration-time curve from time zero to 12 hours. Tinostamustine (EDO-S101) and its metabolites included M2-EDO-S101 and M8-EDO-S101.
Time Frame: Pre-infusion, 0.50, 0.75, 1, 3, 6 hours post-infusion
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Tinostamustine 180 mg/m^2 | Tinostamustine 220 mg/m^2
Number analyzed (Participants) | 2 | 3
h*ng/mL
  EDO-S101 | NA (NA) — Mean and SD was not calculated as data were available for only two participants. | 4887.16 (2052.21)
  M2-EDO-S101: number analyzed (Participants) | 0 | 0
  M8-EDO-S101: number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of tinostamustine up to end of study (up to 6 months)
Description: Safety population included all participants who received tinostamustine.
Groups:
- Tinostamustine (180 mg/m^2): Participants received single dose of 180 mg/m^2 tinostamustine IV injection on Day -1 followed by ASCT on Day 1.
- Tinostamustine (220 mg/m^2): Participants received single dose of 220 mg/m^2 tinostamustine IV injection on Day -1 followed by ASCT on Day 1.
Arm/Group | Tinostamustine (180 mg/m^2) | Tinostamustine (220 mg/m^2)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tinostamustine (180 mg/m^2) (N=3) | Tinostamustine (220 mg/m^2) (N=3)
Pneumonia (Infections and infestations) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tinostamustine (180 mg/m^2) (N=3) | Tinostamustine (220 mg/m^2) (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Anal incontinence (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 2 | 3
Lymphocyte count decreased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 1 | 1
Blood creatinine increased (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0
Thrombosis in device (Product Issues) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 2
Deep vein thrombosis (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Study was early terminated during Phase 1 due to sponsor decision on 17 April 2019 (adverse events limited administration of higher doses required to achieve myeloablative conditioning necessary in this population). Hence, no participants were enrolled in Phase 2 and efficacy analysis were not performed in the both Phase 1 and 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-06-18): https://cdn.clinicaltrials.gov/large-docs/25/NCT03687125/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/25/NCT03687125/SAP_001.pdf